CLINICAL TRIAL: NCT02330614
Title: Is the Personality Relevant in the Choice of Bleaching ?
Brief Title: Personality Bleaching
Acronym: NEOFFI
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof.Eduardo Fernández G., University of Chile
Other Study IDs: 2013-18
Record Dates: First submitted 2014-12-27; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Personality
Keywords: personality; bleaching

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- bleaching patients: Patients who agreed to be bleaching were treated with 10% carbamide peroxide (CP) gel (Whiteness Perfect, FGM) to each subject With verbal instructions for 3 weeks with daily applications of 1 hour according to manufacturers indications , before and after this procedure was applied again the NEO-FFI personality test form, had 30 minutes to answer it.
  Interventions: Other: Bleaching by peroxide carbamide 10%
- Control group: Patients who refused to be bleached were administered the personality test NEO-FFI, had 30 minutes to answer it.
  Interventions: Other: Nothing - control group

INTERVENTIONS:
Other: Bleaching by peroxide carbamide 10% — bleaching were treated with 10% carbamide peroxide (CP) gel (Whiteness Perfect, FGM) to each subject With verbal instructions for 3 weeks with daily applications of 1 hour according to manufacturers indications
  Groups: bleaching patients
Other: Nothing - control group — Only NEO-FFI test , data used as control
  Groups: Control group

SUMMARY:
128 patients between 18 and 76 years who attended the Operative Dentistry Clinic at Dental School, Universidad de Chile, were included in the study. 58 patients were bleaching (experimental group) and 70 patients don't accepted the bleaching procedure (control group) were included in this study and signed a consent form.Experimental group Patients who agreed to be bleaching were treated with 10% carbamide peroxide (CP) gel (Whiteness Perfect, FGM) to each subject With verbal instructions for 3 weeks with daily applications of 1 hour according to manufacturers indications , before and after this procedure was applied again the NEO-FFI personality test form, had 30 minutes to answer it.Control group:Patients who refused to be bleached were administered the personality test NEO-FFI, had 30 minutes to answer it.

DETAILED DESCRIPTION:
Data collection NEO-FFI data was collected in a Microsoft Excel data sheet and analyzed by a psychology that was blind to patient's expectations. According to the answers, each scale might get a score between 0 and 50.

Statistical analysis For comparisons between scales between groups of patients were bleaching and who refused to be bleached Mann Whitney test was used.For each pair of scales it was determined if any one of them predominated over its counterpart by Wilcoxon rank test before and after bleaching . To corroborate the statistical power of this study was calculated post-hoc with the NEO-FFI scores values between the comparisons and showed a high statistical power (0.99) by G-Power software.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in this clinical trial were between 18 and 76 years old and had good general and oral health. Each subject had at least one central incisor with shade A2 or darker, assessed by comparison with a value-oriented shade guide (Vita classical, Vita Zahnfabrik, Bad Säckingen, Germany)

Exclusion Criteria:

* Participants that had undergone previous dental bleaching procedures during orthodontic treatment, or those that were pregnant or lactating women and participants with bruxism habits, were not included in the trial. Additionally, participants with restorations on the labial surfaces of their anterior teeth and non-carious cervical lesions, veneers or full crowns, with gingival recession, spontaneous tooth pain, internal tooth discoloration, and teeth with endodontic treatment or fluorosis were also excluded from this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 128 patients between 18 and 76 years who attended the Operative Dentistry Clinic at Dental School, Universidad de Chile, were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
NEO-FFI score | Baseline / 1 month after

CONTACTS AND LOCATIONS:
Overall Officials: eduardo fernandez, Principal Investigator — University of Chile